CLINICAL TRIAL: NCT01894906
Title: A Controlled, Randomized Study to Assess the Quantitative Mass Transfer of Iron From SFP-containing Hemodialysate Under Varying Conditions of Blood and Dialysate Flow Rates, Dialyzer Membrane Types and Dialysate Bicarbonate Concentrations in CKD-HD Patients.
Brief Title: Quantitative Mass Transfer of SFP-iron From Dialysate to Blood in CKD-HD Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rockwell Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RMTI-SFP-8
Record Dates: First submitted 2013-06-27; First posted 2013-07-10 (Estimated); Results first posted 2015-01-09 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-01

CONDITIONS: Kidney Failure
Keywords: Soluble Ferric Pyrophosphate,; Pharmacokinetics,; Iron, Mass Transfer,; Hemodialysis; chronic therapy;
MeSH Terms: conditions — Renal Insufficiency | interventions — spleen fibrinolytic proteinase (human)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Each subject will receive one control treatment and 5 treatments with SFP added to dialysate. The 5 SFP treatments will encompass 5 different conditions which may impact the intradialytic transfer of iron to the subject: new dialyzer, reused dialyzer, low blood/dialysate flow rate, low machine delivered bicarbonate concentration, and a different synthetic dialysis membrane (PAES).
  Interventions: Other: Placebo
- Soluble Ferric Pyrophosphate (Experimental): Group/ cohort designation: Cellulose dialysis membrane (CT-190)/ Polyamide membrane. Each subject will receive one control treatment and 5 treatments with SFP added to dialysate. The 5 SFP treatments will encompass 5 different conditions which may impact the intradialytic transfer of iron to the subject: new dialyzer, reused dialyzer, low blood/dialysate flow rate, low machine delivered bicarbonate concentration, and a different synthetic dialysis membrane (PAES).
  Interventions: Drug: Soluble Ferric Pyrophosphate

INTERVENTIONS:
Drug: Soluble Ferric Pyrophosphate
  Other Names: SFP
  Arms: Soluble Ferric Pyrophosphate
Other: Placebo
  Arms: Control

SUMMARY:
The purpose of this study is to determine the quantity of iron derived from SFP that is transferred from the dialysate to patients during a single dialysis session. The effects of various conditions which may affect the transfer of iron such as blood and dialysate flow rate, changes in bicarbonate delivery, dialyzer membrane type and the effect of reuse will also be investigated. The absorption and removal of iron from the blood will also be investigated.

DETAILED DESCRIPTION:
* A total of 12 subjects on standard 3X/week hemodialysis will be studied in 2 groups (6 subjects per group)
* 2 primary dialyzer membranes will be studied.:

  * Polyamide Membrane (Gambro Polyflux series: 17R and 21R)
  * Cellulose Triacetate (Baxter CT series: CT-190)
* Each 1-week treatment cycle will include 3 haemodialysis (HD) sessions per subject, including 2 study treatment-HD sessions and 1 non-treatment-HD session per subject. Treatment-HD sessions will be conducted midweek and end-of-week (i.e. Dialysis days 3 and 5 of each week with a 1 day interdialytic interval) to avoid excessive fluid shifts due to the increased UF needed during the non-treatment HD session (conducted at beginning of the week; HD day 1).
* Within each group, each subject will be randomized to 1 of 6 treatment sequences. The treatments to be investigated are: Control; new dialyzer, reused dialyzer, low blood flow/dialysate flow, Low bicarbonate concentration and a different synthetic dialyzer membrane (PAES)
* Blood for a complete serum iron profile over time will be obtained during the new dialyzer (SFP/standard bicarbonate/new dialyzer/ high Qb and Qd) for all subjects. This will necessitate approximately a 24-hour inpatient confinement to obtain blood at specified time intervals after dialysis is completed. Blood for a partial iron profile will be collected during the dialysis sessions at all other dialysis sessions.
* Each of the 6 enrolled subjects per dialyzer membrane type will be assigned to a different sequence of treatments to help ensure that the treatment sequence does not affect the analysis (Note: the first dialysis sessions of each of the 3 study weeks, i.e. HD1, HD4 and HD7, are non-study related sessions during which no study procedures are performed except for adverse event collection.
* Patients should not be receiving any of the following medications from screening through the end of the study:

  * Oral iron preparations, including multivitamin supplements containing iron
  * Intravenous iron preparations
* Doses of ESA's should not be changed from screening to the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subject ≥ 18 years of age undergoing chronic hemodialysis for chronic kidney disease (CKD) for at least 3 months, expected to remain on hemodialysis and be able to complete the study.
2. Screening Hgb ≥ 9.5 g/dL.
3. Screening transferrin saturation % (TSAT) ≥ 15% to ≤ 45%.
4. Screening serum ferritin ≥ 200 to ≤ 1200 µg/L.
5. Subject's standard dialyzer membrane is one of the 2 types, i.e. Baxter CT-190 or Gambro 17R or 21R.
6. The subject uses a reprocessed dialyzer for standard HD treatments.
7. Prescribed dialysis 3X/week.
8. Minimally adequate measured dialysis dose defined as URR (urea reduction ratio) ≥ 65%, or single-pool Kt/V (dialyzer clearance of urea multiplied by dialysis time, divided by patient's total body water) ≥ 1.2, or KIDt/V (online dialyzer clearance measured using ionic dialysance multiplied by dialysis time, divided by patients total body water) ≥ 1.2.
9. Stable dialyzer blood flow rate that is generally ≥ 350 mL/min and acceptable to the Investigator.
10. Stable dialysate flow rate that is generally ≥ 600 mL/min and acceptable to the Investigator.
11. Vascular access for dialysis that will be used upon enrollment with stable function in the judgment of the Investigator.
12. Female subjects must be either amenorrheic for ≥ 1 year or agree to not become pregnant by continuous use of an effective birth control method acceptable to the Investigator for the duration of their participation in the study.
13. Must be willing and able to provide written informed consent directly or through their authorized representative.

Exclusion Criteria:

1. Subject has a living kidney donor identified or living-donor kidney transplant scheduled during study participation. (Note: Patients awaiting deceased-donor transplant need not be excluded.)
2. Vascular access for hemodialysis is a femoral catheter.
3. Known active bleeding from any site other than AV fistula or graft (e.g., gastrointestinal, hemorrhoidal, nasal, pulmonary, etc.).
4. Scheduled surgery during the study.
5. RBC or whole blood transfusion within 4 weeks prior to Screening.
6. Hospitalization in the month prior to Screening (except for vascular access surgery) that, in the opinion of the Investigator, confers a significant risk of hospitalization during the course of this study.
7. Evidence of current malignancy involving a site other than skin (except any melanoma, which renders the patient non-eligible).
8. History of drug or alcohol abuse within the last 6 months.
9. Regularly requiring hemodialysis more than three times per week.
10. Noncompliance with dialysis regimen in the opinion of the Investigator.
11. Pregnancy or intention to become pregnant before completing all study drug treatment.
12. Known ongoing inflammatory disorder (other than CKD), such as systemic lupus erythematosus, rheumatoid arthritis, or other collagen-vascular disease undergoing a disease flare.
13. Any current febrile illness (e.g., oral temperature > 100.4°F, 38°C). (The patient may subsequently become eligible at least 1 week after resolution of the illness).
14. Known active bacterial, tuberculosis, fungal, viral, or parasitic infection requiring anti-microbial therapy or anticipated to require anti-microbial therapy during the patient's participation in this study.
15. Occult tuberculosis requiring prophylactic treatment with anti-tubercular drug(s) that overlaps with the patient's participation in this study.
16. Known positive status for hepatitis B surface antigen (hepatitis B testing is not required as part of this protocol).
17. Known human immunodeficiency virus (HIV) infection (HIV testing is not required as part of this protocol).
18. Cirrhosis of the liver based on histological criteria or clinical criteria (i.e., presence of ascites, esophageal varices, multiple spider nevi, or history of hepatic encephalopathy).
19. Active hepatitis with ALT and/or AST levels consistently greater than twice the upper limit of normal at any time during the two months prior to enrollment.
20. Participation in a study of an investigational drug or device within 30 days prior to randomization in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond D Pratt, MC FACP, Study Director — Rockwell Medical Inc
Locations (1):
- Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 19 patients were screened and 12 total patients were enrolled. Each patient participated in each of the 6 treatment periods.
Groups:
- Baxter CT-190 (Group 1: Cellulose Triacetate Membrane); Gambro 17R/21R (Group 2: Polyamide Membrane): Enrolled subjects were assigned to 1 of 2 groups based on the type of dialyzer membrane used by each subject at Screening: Baxter CT-190 (Group 1; N = 6; cellulose triacetate membrane) or Gambro 17R/21R (Group 2; N = 6; polyamide membrane). Within each dialyzer membrane group, each subject received one control treatment and 5 treatments with SFP added to dialysate.
Period: Overall Study
Arm/Group | Baxter CT-190 (Group 1: Cellulose Triacetate Membrane) | Gambro 17R/21R (Group 2: Polyamide Membrane)
Started | 6 | 6
Treatment A | 6 | 6
Treatment B | 6 | 6
Treatment C | 6 | 6
Treatment D | 6 | 6
Treatment E | 6 | 6
Treatment F | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No prospective calculations of statistical power were made. The sample size of 12 subjects (N = 6 for each of 2 dialysis membrane groups) was selected to provide information on safety and to provide preliminary data for assessing the variance of iron delivery under different, pre-specified dialysis conditions.
Groups:
- Total: Total of all reporting groups
Arm/Group | Baxter CT-190 (Group 1: Cellulose Triacetate Membrane) | Gambro 17R/21R (Group 2: Polyamide Membrane). | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (14.73) | 52.8 (8.89) | 52.3 (11.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.425 (6.1611) | 28.332 (6.6425) | 27.378 (6.1888)

OUTCOME MEASURES:

1. Secondary Outcome: To Compare the Amount of SFP-derived Iron Administered Under Various Treatment Conditions to the Reference HD
Description: To compare the amount of SFP-derived iron administered under various treatment conditions to the reference HD (Treatment B: SFP, new membrane, high Qb/Qd, 37 mEq bicarbonate): Dialyzer reuse, Low machine bicarbonate delivery, Polyarylethersulfone (PAES) membrane, and Low Qb/Qd.Iron concentration in timed dialysate collections will be analyzed. Expended dialysate over the intervals of 0.5, 1, 2 ,3 and 4 hours will be collected and measured. Aliquots will be analyzed for iron content. The mean cumulative net iron delivery will be reported.
Time Frame: one dialysis session (approximately 4 hours)
Population: For this preliminary and explorative study, no prospective calculations of statistical power were made; statistics were descriptive only. All subjects were included in the calculation of all study outcomes.
Measure: Mean (Standard Deviation); unit: microgram
Groups:
- Control: Enrolled subjects were assigned to 1 of 2 groups based on the type of dialyzer membrane used by each subject at Screening: Baxter CT-190 (Group 1; N = 6; cellulose triacetate membrane) or Gambro 17R/21R (Group 2; N = 6; polyamide membrane). Within each dialyzer membrane group, each subject received one control treatment and 5 treatments with SFP added to dialysate. Treatment A was one dialysis session without SFP added to the bicarbonate, with standard bicarbonate concentration, blood flow rate, dialysis flow rate, and new dialyzer.
- Treatment B: Enrolled subjects were assigned to 1 of 2 groups based on the type of dialyzer membrane used by each subject at Screening: Baxter CT-190 (Group 1; N = 6; cellulose triacetate membrane) or Gambro 17R/21R (Group 2; N = 6; polyamide membrane). Within each dialyzer membrane group, each subject received one control treatment and 5 treatments with SFP added to dialysate. Treatment B was one dialysis session with SFP added to the bicarbonate, with standard bicarbonate concentration, blood flow rate, dialysis flow rate, and new dialyzer.
- Treatment C: Enrolled subjects were assigned to 1 of 2 groups based on the type of dialyzer membrane used by each subject at Screening: Baxter CT-190 (Group 1; N = 6; cellulose triacetate membrane) or Gambro 17R/21R (Group 2; N = 6; polyamide membrane). Within each dialyzer membrane group, each subject received one control treatment and 5 treatments with SFP added to dialysate. Treatment C was one dialysis session with SFP added to the bicarbonate, with standard bicarbonate concentration, blood flow rate, dialysis flow rate, and re-used dialyzer.
- Treatment D: Enrolled subjects were assigned to 1 of 2 groups based on the type of dialyzer membrane used by each subject at Screening: Baxter CT-190 (Group 1; N = 6; cellulose triacetate membrane) or Gambro 17R/21R (Group 2; N = 6; polyamide membrane). Within each dialyzer membrane group, each subject received one control treatment and 5 treatments with SFP added to dialysate. Treatment D was one dialysis session with SFP added to the bicarbonate, with low bicarbonate concentration, blood flow rate, dialysis flow rate, and new dialyzer.
- Treatment E: Enrolled subjects were assigned to 1 of 2 groups based on the type of dialyzer membrane used by each subject at Screening: Baxter CT-190 (Group 1; N = 6; cellulose triacetate membrane) or Gambro 17R/21R (Group 2; N = 6; polyamide membrane). Within each dialyzer membrane group, each subject received one control treatment and 5 treatments with SFP added to dialysate. Treatment E was one dialysis session with SFP added to the bicarbonate, with standard bicarbonate concentration, low blood flow rate, low dialysis flow rate, and new dialyzer.
- Treatment F: Enrolled subjects were assigned to 1 of 2 groups based on the type of dialyzer membrane used by each subject at Screening: Baxter CT-190 (Group 1; N = 6; cellulose triacetate membrane) or Gambro 17R/21R (Group 2; N = 6; polyamide membrane). Within each dialyzer membrane group, each subject received one control treatment and 5 treatments with SFP added to dialysate. Treatment B was one dialysis session with SFP added to the bicarbonate, with standard bicarbonate concentration, blood flow rate, dialysis flow rate, and new Gambro 17R/21R PAES membrane dialyzer.
Arm/Group | Control | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12
microgram | -18.5 (175) | 692 (1010) | 578 (1380) | 587 (994) | 130 (594) | 350 (1940)

2. Secondary Outcome: Pharmacokinetics of Serum Iron and Exploratory Modeling
Description: The serum Total Iron, Transferrin Bound Iron (TBI) and Non-transferrin Bound Iron (NTBI) pharmacokinetic parameters (baseline corrected and total) will be listed and summarized for each membrane group and overall. The mean serum total iron, TBI, NTBI, unsaturation iron binding capacity (UIBC) and total iron binding capacity (TIBC) concentrations at baseline (BL), end-of-treatment, and the change from BL will be listed for each group (Baxter and Gambro Polyflux), measured from the reference HD (Treatment B: SFP, new membrane, high Qb/Qd, 37 mEq bicarbonate).
Time Frame: one dialysis session (approximately 4 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microgram/dL
Groups:
- Baxter CT-190; Gambro Polyflux: Enrolled subjects were assigned to 1 of 2 groups based on the type of dialyzer membrane used by each subject at Screening: Baxter CT-190 (Group 1; N = 6; cellulose triacetate membrane) or Gambro 17R/21R (Group 2; N = 6; polyamide membrane).
- Baxter and Gambro Combined: Enrolled subjects were assigned to 1 of 2 groups based on the type of dialyzer membrane used by each subject at Screening: Baxter CT-190 (Group 1; N = 6; cellulose triacetate membrane) or Gambro 17R/21R (Group 2; N = 6; polyamide membrane). This category includes the combined results of both groups.
Arm/Group | Baxter CT-190 | Gambro Polyflux | Baxter and Gambro Combined
Number analyzed (Participants) | 6 | 6 | 12
microgram/dL
  Baseline TIBC | 244.7 (49.31) | 221.7 (52.88) | 233.2 (50.21)
  End-of Treatment TIBC | 247.2 (39.83) | 233.5 (61.40) | 240.3 (49.85)
  TIBC Change from BL to EoT | 2.5 (41.95) | 11.8 (14.50) | 7.2 (30.32)

3. Primary Outcome: Net Iron Delivery From SFP Via the Dialysate
Description: To measure the SFP-derived total iron from the reference HD (Treatment B: SFP, new membrane, high Qb/Qd, 37 mEq bicarbonate). Expended dialysate over the intervals of 0.5, 1, 2 ,3 and 4 hours will be collected and measured. Aliquots will be analyzed for iron content. The mean cumulative net iron delivery will be reported.
Time Frame: one dialysis session (approximately 4 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microgram
Arm/Group | Treatment B
Number analyzed (Participants) | 12
microgram | 692 (1010)

4. Secondary Outcome: Dialysate InFlow Iron Concentration
Description: Dialysate inflow iron concentration was calculated for each treatment group at t = 0, 0.5, 1, 2, 3, and 4 hours.
Time Frame: 4 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micrograms/L
Arm/Group | Control | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12
micrograms/L
  t = 0 hours | 12.5 (43.3) | 0 (0) | 0 (0) | 1.9 (6.58) | 0 (0) | 0 (0)
  t = 0.5 hours | 0 (0) | 71 (6.87) | 74.1 (9.44) | 63.3 (5.5) | 54.7 (4.61) | 64.4 (14)
  t = 1 hour | 0 (0) | 74 (2.53) | 76.3 (7.46) | 63.9 (5.12) | 56.6 (5.32) | 69.2 (13.3)
  t = 2 hours | 0.925 (3.2) | 74.4 (2.66) | 75.9 (7.73) | 64.4 (5.37) | 58.2 (7.57) | 68.5 (14)
  t = 3 hours | 0 (0) | 71.9 (6.98) | 76.8 (8.75) | 64.8 (5.84) | 57.7 (8.36) | 69.1 (12.2)
  t = 4 hours | 0 (0) | 73.6 (3.4) | 73.3 (5.74) | 63.7 (6.64) | 56.1 (4.8) | 69.3 (14.6)

5. Secondary Outcome: Dialysate OutFlow Iron Concentration
Description: Dialysate outflow iron concentration was calculated for each treatment group at t = 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, and 4 hours.
Time Frame: 4 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micrograms/L
Arm/Group | Control | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12
micrograms/L
  t = 0.25 hours | 0.643 (2.23) | 68.6 (8.15) | 73.1 (11.2) | 61.8 (6.7) | 53 (7.16) | 66.2 (9.19)
  t = 0.5 hours | 3.21 (11.1) | 68.4 (8.22) | 74.1 (11.1) | 62.2 (7.62) | 54.3 (8.36) | 65.6 (9.85)
  t = 0.75 hours | 0 (0) | 81.8 (25.9) | 74.9 (11.6) | 62 (8.61) | 50.4 (17.4) | 64.8 (11.7)
  t = 1 hour | 0 (0) | 64.4 (22.1) | 74.1 (13.3) | 61.6 (9.1) | 53.5 (8.41) | 68.5 (12.2)
  t = 1.5 hours | 0 (0) | 74.2 (5.04) | 73.6 (12.6) | 61.8 (8.2) | 53.8 (9.09) | 65.4 (9.44)
  t = 2 hours | 0 (0) | 70.9 (8.56) | 71.9 (17.4) | 63.4 (6.99) | 57.2 (6.27) | 65.3 (10.8)
  t = 2.5 hours | 1.74 (6.03) | 70.6 (8.26) | 75 (15) | 58.1 (12) | 55.4 (7.65) | 65.8 (10.7)
  t = 3 hours | 0 (0) | 77.9 (17.8) | 75.6 (10.4) | 60.6 (7.21) | 55.2 (8.42) | 64.3 (13.5)
  t = 3.5 hours | 0 (0) | 74 (10.5) | 71.6 (13.7) | 56.5 (3.1) | 53.3 (4.75) | 71.4 (8.62)
  t = 4 hours | 0 (0) | 72.4 (6.03) | 76.5 (13.1) | 60.8 (8.81) | 54.4 (9.08) | 66.3 (12.6)

ADVERSE EVENTS:
Arm/Group | Control | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 2/12 | 2/12 | 1/12 | 2/12 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=12) | Treatment B (N=12) | Treatment C (N=12) | Treatment D (N=12) | Treatment E (N=12) | Treatment F (N=12)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Total iron, TBI, NTBI, and UIBC could not be measured because the ferrozine assay for total iron and transferrin-bound iron was unreliable due to the presence of heparin in the samples, which caused the formation of fibrin strands.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less